CLINICAL TRIAL: NCT06181786
Title: A Randomized, Double-Blind, Placebo-controlled, Single and Multiple Ascending Dose Phase 1 Clinical Study to Evaluate Safety, Tolerability, and Pharmacokinetics of NAV-240 in Healthy Volunteers
Brief Title: Study of NAV-240 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Navigator Medicines, Inc. (Industry)
Collaborators: IMBiologics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IMB101-CR-01
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: Pharmacokinetics; IMB-101; OX40L/TNF bispecific antibody; NAV-240

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Ascending Doses (SAD) of NAV-240 IV (Experimental): Single intravenous (IV) administration of ascending dose levels of NAV-240
  Interventions: Drug: NAV-240
- Single Doses of Placebo (Placebo Comparator): Single intravenous (IV) administration of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NAV-240 — Intravenous administration of NAV-240
  Arms: Single Ascending Doses (SAD) of NAV-240 IV
Drug: Placebo — Intravenous administration of matching placebo for NAV-240
  Arms: Single Doses of Placebo

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of intravenous (IV) doses of NAV-240 in healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

1. The participant is 18 to 55 years of age, inclusive, at screening.
2. The participant has a BMI of 18.5 to ≤ 32 kg/m^2 at screening.
3. The participant is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings not clinically significant at screening.
4. Female participants of childbearing potential must use at least 1 form of highly effective methods of birth control from screening until at least 90 days after last study drug dose; OR be surgically sterile OR be postmenopausal. All female participants of childbearing potential must have a negative pregnancy test at screening and before the first dose of study drug. Female participants must also agree to refrain from egg donation during the study and for at least 90 days after study drug dosing.
5. Male participants must agree to use a condom when sexually active with a female partner of childbearing potential during the study and for at least 90 days after study drug dosing (OR be surgically sterile; OR agree to practice abstinence during the study and for at least 90 days after study drug dosing).
6. The participant agrees to comply with all protocol requirements.
7. The participant is able to provide written informed consent.

Key Exclusion Criteria:

1. The participant has any significant acute or chronic medical illness that, in the opinion of the investigator, would impact the participant's ability to complete all study requirements or that might impact the assessment of study data; or the participant has had a clinically significant illness within 30 days prior to study drug dosing per investigator discretion.
2. The participant has a positive COVID-19 molecular diagnostic test result at screening or prior to study drug dosing; or the participant has known or suspected current sequelae from a prior episode of COVID-19.
3. The participant has had major surgery, as determined by the investigator, within 12 weeks prior to study drug dosing.
4. The participant has any of the following prior to study drug dosing:

   • Systolic blood pressure >140 mmHg and/or diastolic blood pressure >90 mmHg.
5. The participant has any of the following on 12-lead ECG prior to study drug dosing, confirmed by repeat:

   * Heart rate <40 or >100 beats per minute.
   * PR interval >220 milliseconds (ms).
   * QRS width >120 ms.
   * QTcF >=450 ms (male) or >=470 ms (female).
6. The participant has any of the following clinical laboratory results at screening, confirmed by repeat:

   * WBCs, lymphocytes, or neutrophil counts outside site acceptable ranges per site SOPs.
   * eGFR < 60 mL/min/1.73m^2 (the CKD-EPI formula)
   * ALT or AST >2*ULN
   * Total bilirubin >2*ULN
7. The participant has a positive test result for HBsAg, anti-HBcAb, hepatitis C virus antibody, or HIV types 1 or 2 antibodies at screening.
8. The participant has a history of TB, active TB, or a positive Quantiferon-TB Gold Plus (QFT-Plus) test at screening.
9. The participant has received any vaccine or used any prescription or over the-counter medications (except acetaminophen [up to 2 g per day]), including herbal or nutritional supplements, within 14 days prior to study drug dosing.
10. The participant has received biologic agents within the 3 months prior to study drug dosing, or 5 half-lives, whichever is greater. Participants with a prior history of anti-TNFα exposure will be excluded.
11. The participant is a smoker or has regularly used nicotine or nicotine-containing products within 3 months prior to study drug dosing.
12. History of drug abuse within 1 year prior to screening.
13. The participant has a positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking) at screening or prior to study drug dosing.
14. The participant has donated blood or blood products >500 mL within 30 days prior to study drug dosing.
15. The participant has a history of hypersensitivity to vaccines, the study drug, or to drugs of similar chemical classes including allergy to drug or its excipients.
16. Any reason which, in the opinion of the Investigator, would prevent the participant from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From the dose of study drug on Day 1 up to Day 71
  TEAEs are defined as events that started after the first dose of study treatment or events that presented prior to the first dose of study drug but increased in severity after the first dose based on preferred term, including clinically relevant abnormal laboratory findings.
  SAEs are defined as any event that either results in death, is immediately life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of NAV-240 | From Day 1 prior to the first dose of study drug up to Day 71
Time to Maximum Serum Concentration (Tmax) of NAV-240 | From Day 1 prior to the first dose of study drug up to Day 71
Area Under the Serum Concentration-Time Curve From Time Zero to 336 hours post-dose (AUC0-336) of NAV-240 | From Day 1 prior to the first dose of study drug up to Day 71
Area Under the Serum Concentration-Time Curve from Time Zero to the Concentration at a given Time Point (AUC0-t) of NAV-240 | From Day 1 prior to the first dose of study drug up to Day 71
Area Under the Serum Concentration-Time Curve from Time Zero to Infinity (AUC0-inf) of NAV-240 | From Day 1 prior to the first dose of study drug up to Day 71
Serum Elimination Half-life (t1/2) of NAV-240 | From Day 1 prior to the first dose of study drug up to Day 71
Terminal Elimination Rate Constant (λz) of NAV-240 | From Day 1 prior to the first dose of study drug up to Day 71
Apparent Total Body Clearance (CL) of NAV-240 | From Day 1 prior to the first dose of study drug up to Day 71
Apparent Volume of Distribution (Vz) of NAV-240 | From Day 1 prior to the first dose of study drug up to Day 71
Trough Serum Concentration (Ctrough) of NAV-240 | From Day 1 prior to the first dose of study drug up to Day 71
Incidence of Presence of Antidrug Antibodies (ADAs) | From the first dose of study drug up to Day 71
  The formation of ADAs against NAV-240 as assessed in blood samples. Proportion of participants with positive or negative results for ADAs.
ADA Titers in Participants with Positive ADA | From the first dose of study drug up to Day 71

CONTACTS AND LOCATIONS:
Overall Officials: Dana McClintock, MD, Study Director — Navigator Medicines, Inc.
Locations (1):
- Syneos Health, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No